CLINICAL TRIAL: NCT00931060
Title: Effects of Branched-Chain Amino Acids on Muscle Ammonia Metabolism in Patients With Cirrhosis and Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Gitte Dam, PET Centre. Aarhus University Hospital.
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 15580
Record Dates: First submitted 2009-06-30; First posted 2009-07-02 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Liver Diseases; Hepatic Encephalopathy; Hepatic Insufficiency
Keywords: Ammonia; Citric acid cycle; Branched Chain Amino Acids
MeSH Terms: conditions — Liver Diseases; Hepatic Encephalopathy; Hepatic Insufficiency | interventions — Amino Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Branched chain amino acids (Experimental): Patients with cirrhosis. Healthy subjects age and sex matched
  Interventions: Dietary Supplement: Branched chain amino acids

INTERVENTIONS:
Dietary Supplement: Branched chain amino acids — Branched chain amino acids 0.45g/kg BW. Oral supplement. Administered once on study day

SUMMARY:
The purpose of this study is to determine whether Branched chain Amino Acids enhances the uptake of ammonia in muscle tissue.

DETAILED DESCRIPTION:
Branched-chain amino acids (BCAA; leucine, valine, isoleucine) are used to prevent hepatic encephalopathy in cirrhotic patients. The main effect of BCAAs is believed to take place in muscles where BCAAs provide carbon-skeletons for the TCA-cycle. This enhances the conversion of alfa-ketoglutarate to ammonia via glutamine.

We intend to study the effect of oral administered BCAA on the metabolism of ammonia and amino acids across the leg-muscles by means of catheters inserted into the femoral artery (A) and vein (V). Muscle blood flow (F; L/min) will be determined by constant infusion of indocyanine green and indicator dilution principle. Arterial blood flow and A and V concentrations of ammonia and amino acids will be measured before an oral load of BCAA (0.45 g BCAA/kg body weight) and after 1 and 3 hours. The metabolism of ammonia will also be estimated by means of 13N-NH3 PET scans.

Hypothesis: BCAA increases the uptake of ammonia in muscle tissue and lowers arterial ammonia.

ELIGIBILITY:
Inclusion Criteria:

* 18 patients with liver cirrhosis
* 6 healthy subjects age and sex matched

Exclusion Criteria:

* Non-treated diabetes
* Pregnancy/breast-feeding

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
arterial ammonia concentration | 1 and 3 hours

SECONDARY OUTCOMES:
muscle ammonia metabolism | 1 hour and 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Keiding, MD, Study Chair — PET Centre and Medical department V, Aarhus Sygehus, Aarhus University Hospital